CLINICAL TRIAL: NCT02730494
Title: Study Evaluating the Optimal Dosage for Equivalence Between a Tablet and Capsule Dosage Form of an Intravaginal Treatment With Total Freeze-dried Culture of Lcr Regenerans® (Lactobacillus Rhamnosus Lcr35®) on Vaginal Flora Colonisation in Healthy Women.
Brief Title: Study Evaluating the Optimal Dosage for Equivalence Between Lcr Regenerans® Capsules and Tablets (Lactobacillus Rhamnosus Lcr35®) on the Vaginal Flora Colonisation
Acronym: COMPRIGEL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biose (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PRO_2014-01; 2014-001746-21 (EudraCT Number)
Record Dates: First submitted 2016-04-01; First posted 2016-04-06 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Candidiasis, Vulvovaginal
Keywords: mycosis; Candidiasis; Lcr35®; Lcr Regenerans®
MeSH Terms: conditions — Candidiasis, Vulvovaginal; Mycoses; Candidiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Lcr Regenerans® vaginal capsule (Active Comparator): Name: Lcr Regenerans® containing at least 10e7 CFU per intravaginal capsule. 1 vaginal capsule per day
  Interventions: Device: Lcr Regenerans® vaginal capsules
- Lcr Regenerans® vaginal tablet every 3 days (Experimental): Lcr Regenerans® containing at least 10e7 CFU per intravaginal table. One vaginal tablet every 3 days
  Interventions: Device: Lcr Regenerans® vaginal tablet
- Lcr Regenerans® vaginal tablet every 4 days (Experimental): Lcr Regenerans® containing at least 10e7 CFU per intravaginal table. One vaginal tablet every 4 days
  Interventions: Device: Lcr Regenerans® vaginal tablet
- Lcr Regenerans® vaginal tablet every 5 days (Experimental): Lcr Regenerans® containing at least 10e7 CFU per intravaginal table. One vaginal tablet every 5 days
  Interventions: Device: Lcr Regenerans® vaginal tablet

INTERVENTIONS:
Device: Lcr Regenerans® vaginal capsules
  Other Names: GYNOPHILUS Capsules
  Arms: Lcr Regenerans® vaginal capsule
Device: Lcr Regenerans® vaginal tablet
  Other Names: GYNOPHILUS Tablet
  Arms: Lcr Regenerans® vaginal tablet every 3 days; Lcr Regenerans® vaginal tablet every 4 days; Lcr Regenerans® vaginal tablet every 5 days

SUMMARY:
The primary objective of this study is to study the vaginal flora colonisation equivalence between the tablet and capsule dosage forms of a treatment with Lcr Regenerans® between D0 (V1) and Dend of treatment.

DETAILED DESCRIPTION:
The healthy vaginal microbiota is mainly colonised by strains of Lactobacillus which play an important role in defence against vaginal infections. The intravaginal use of probiotic strains stimulating the recolonisation of the endogenous vaginal microbiota and capable of inhibiting the growth of pathogens such as Candida albicans appears to be an interesting alternative to prevent recurrences of VVC. Recently, longitudinal studies have revealed that the vaginal microbiota is relatively stable and that the main cause of disturbance to the stability of the vaginal microbiota is over short menstruation periods. However, the use of antimicrobial agents induces severe disturbances with disappearance of certain endogenous species over several weeks. These results suggest that antimicrobial treatments severely affect the vaginal flora and that probiotics are therefore recommended to help re-establish a vaginal microbiota after this treatment.

For this, a sufficient direct local supply must be provided. The general data from studying the vaginal microbiota reveal that in the healthy woman, the concentration of Lactobacilli is greater than or equal to 107 CFU/ml of vaginal secretion. During capsule administration, all the Lactobacilli are immediately released into the vaginal cavity. The natural vaginal secretions, estimated to be an average of 0.51 ml/day, result in daily elimination of around 107 to 108 CFU and therefore generates very rapid elimination of this supply which requires daily administrations.

The objective of this clinical trial is to prove that the two dosage forms, capsule administered daily and tablet administered at a certain dosage, enable equivalent local provision of a concentration which is greater than or equal to 10e7 CFU (this concentration ensures the establishment of a sufficiently large bacterial population to enable efficacy of the product).

Therefore, the optimal dosage of the Lcr Regenerans® tablet to be administered and which will be equivalent to the daily administration of the Lcr Regenerans® capsule will be determined during this trial. To do this, 3 different dosages of the Lcr Regenerans® tablet, corresponding to or encompassing the time during which the tablet provides continuous release and presence of the strain in the in vitro model, will be compared to that of the Lcr Regenerans® capsule. For this reason, the frequencies of administration for the Lcr Regenerans® tablet will be 3, 4 or 5 days.

ELIGIBILITY:
Inclusion Criteria:

Relating to the condition:

* Clinically healthy women

Relating to the population:

* Adult women
* Women of child-bearing age: with a negative urine pregnancy test and using a method of contraception deemed effective by the investigator(excluding spermicides) throughout the trial
* Women who can be treated with the study product immediately after the inclusion visit for a duration of 21 consecutive days without interruption by her next menstrual period.
* Women who can speak and read French and having been informed about the study and having voluntarily signed an Informed Consent Form
* Women registered with a social insurance scheme

Exclusion Criteria:

* Relating to the condition or the gynaecological field:
* Presence of a presumed or proven gynaecological bacterial or viral infection, whether treated or not during the month preceding inclusion.
* Presence of an existing gynaecological condition that could interfere with the assessment of the trial treatment (severe cervical dysplasia or carcinoma in situ, invasive carcinoma, intra-epithelial cervical neoplasia, squamous intra-epithelial lesions etc.)

Relating to the treatments:

* Systemic antifungals or antibiotics during the month preceding the inclusion visit.
* Use of probiotics (see list in 16.2) during the month preceding the inclusion visit.
* Use of prebiotics (acidifying agents) - (see list in 16.2) during the 15 days preceding the inclusion visit.
* Allergy to one of the active ingredients or one of the excipients in the products.

Relating to the population:

* Women unable to comply with the constraints of the protocol.
* Breastfeeding women.
* Post-menopausal women.
* Women whose menstrual bleeding lasts longer than 8 days per month.
* Women having participated in a clinical study in the 3 months preceding inclusion in this protocol.
* Women with a severe acute or chronic condition deemed by the investigator as being incompatible with participation in the trial or a serious infection which could be life-threatening in the short term.
* Immunosuppressed women.
* Women with a previous condition which, according to the investigator, is likely to interfere with the study results or expose the female volunteer to additional risk.
* Women with linguistic (not speaking or writing French) or psychological inability to understand and sign the informed consent form.
* Women deprived of her liberty through an administrative or judicial decision or subject to a guardianship order.
* Women likely not to comply with the treatment.
* Women who cannot be contacted in the case of emergency.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-07; Primary Completion 2016-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Measure the vaginal flora equivalence between the tablet and the capsule dosage forms of a treatment with Lcr Regenerans® between D0 (V1) and Dend of treatment. | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Yann Dr LENGLET, Principal Investigator — Hospital center Jacques LACARIN of VICHY
Locations (1):
- BIOSE, Aurillac, France